CLINICAL TRIAL: NCT05377736
Title: Thyroid Nodule Gene Sequencing in a Danish Population - a Pilot Study
Brief Title: Thyroid Nodule Gene Sequencing in a Danish Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kristine Zøylner Rubeck, Principal investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Thy-sec-da 032022
Record Dates: First submitted 2022-03-15; First posted 2022-05-17 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Nodule (Diagnosis); Thyroid Cancer
MeSH Terms: conditions — Thyroid Nodule; Disease; Thyroid Neoplasms | interventions — Molecular Docking Simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Molecular testing (Experimental): Descriptive and explorative study including identical molecular analyses applied to all included patients
  Interventions: Genetic: Molecular analyses

INTERVENTIONS:
Genetic: Molecular analyses — Collect thyroid tissue for molecular analysis from the histological specimen collected by routine surgery

SUMMARY:
This pilot study aims at describing the prevalence and distribution of molecular alterations in thyroid nodules of benign and malignant origin at the level of DNA and RNA in a Danish population.

Patients with thyroid nodules suspected of malignancy is included prospectively.

Tissue samples are collected for molecular analyses form surgical specimens and bloodsamples, and preoperative clincial features are registered.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid nodule >1.5 cm
* BSRTC: IV, V, og VI

Exclusion Criteria:

* No surgical specimen available
* Purely cystic nodules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
DNA alterations | Two years
  Whole genome sequencing by next generation sequencing
RNA alterations | Two years
  Total RNA sequencing including circular RNA, micro RNA and messenger RNA
DNA methylation | Two years
  Whole Genome Bisulfite Sequencing
Circulating tumor DNA | Two years
  Whole genome sequencing of leucocyt DNA and circularing DNA

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Z Swan, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus Universityhospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD will be in accordance with Danish legislation and regulations within the area